CLINICAL TRIAL: NCT05252234
Title: Post SARS-Cov-2 Disease Anesthesia Events
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Amr M Hilal Abdou, Assistant professor, Ain Shams University
Other Study IDs: R 191/2021
Record Dates: First submitted 2022-02-19; First posted 2022-02-23 (Actual); Last update posted 2022-03-15 (Actual); Status verified 2022-03

CONDITIONS: Intraoperative Hypertension; Pain Threshold; Postoperative Pain; Postoperative Hypoxemia
Keywords: SARS-Cov-2; Anesthesia
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group 1: Patients undergoing elective surgeries with past history of COVID-19 infection during the past six months
  Interventions: Other: Observation of hemodynamic status and post operative pain

INTERVENTIONS:
Other: Observation of hemodynamic status and post operative pain — No intervention

SUMMARY:
Estimating and recording the rate of occurrence of pulmonary and cardiovascular complications during the perioperative period in patients with past covid infection

ELIGIBILITY:
Inclusion Criteria:

* all patients above 18 years with past history of covid-19 during past 6 months undergoing surgery

Exclusion Criteria:

* hemodynamically unstable Patients requiring oxygen therapy

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Above 18 years undergoing surgery with past history of covid-19
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2022-04-01 (Estimated); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-09-30 (Estimated)

PRIMARY OUTCOMES:
Rate of occurrence of pulmonary and cardiovascular complications | 24 hours
  Measure all vital data and postoperative status

CONTACTS AND LOCATIONS:
Overall Officials: Fathy Tash, MD, Study Chair — Ain Shams University
Locations (1):
- Faculty of medicine, Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 6 months